CLINICAL TRIAL: NCT03205345
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Emricasan, an Oral Caspase Inhibitor, in Subjects With Decompensated Non-Alcoholic Steatohepatitis (NASH) Cirrhosis
Brief Title: Emricasan, a Caspase Inhibitor, for Treatment of Subjects With Decompensated NASH Cirrhosis
Acronym: ENCORE-LF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IDN-6556-17
Record Dates: First submitted 2017-06-20; First posted 2017-07-02 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Decompensated Cirrhosis
Keywords: Cirrhosis; NASH Cirrhosis; Decompensated NASH cirrhosis; Cirrhosis, Liver; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Fibrosis; Liver Cirrhosis; Non-alcoholic Fatty Liver Disease | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study drug will be double-blind with matching placebo. Emricasan at 25 mg or 5 mg or matching placebo will be administered orally twice a day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Emricasan (25 mg) (Active Comparator): Emricasan 25 mg
  Interventions: Drug: Emricasan (25 mg)
- Emricasan (5 mg) (Active Comparator): Emricasan 5mg
  Interventions: Drug: Emricasan (5 mg)
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emricasan (25 mg) — 25 mg emricasan
  Other Names: IDN-6556
  Arms: Emricasan (25 mg)
Drug: Emricasan (5 mg) — 5 mg emricasan
  Other Names: IDN-6556
  Arms: Emricasan (5 mg)
Drug: Placebo — Matching Placebo
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of emricasan in improving event-free survival based on a composite clinical endpoint (where all-cause mortality, new decompensation events, and MELD score progression are events) in subjects with decompensated NASH cirrhosis.

DETAILED DESCRIPTION:
The study treatment duration will be at least 48 weeks with study visits every 4 weeks up to Week 48 and every 8 weeks after Week 48. All subjects will continue treatment until the last subject in the study reaches 48 weeks in the study. At least 30% of subjects randomized should have baseline MELD score ≥15 and ≤20.

For each subject, the study will consist of:

* Screening period of up to 4 weeks
* Randomized, double-blind treatment period of at least 48 weeks
* A follow-up visit 2 weeks after completion of study drug treatment

The duration of each subject's participation will be at least 54 weeks for those completing the entire study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subjects 18 years or older, able to provide written informed consent and able to understand and willing to comply with the requirements of the study.
2. Cirrhosis due to NASH with exclusion of other causes of cirrhosis (e.g. chronic viral hepatitis, alcoholic liver disease, etc.)
3. At least one of the following: a) history of variceal hemorrhage (more than 3 months prior to day 1) documented on endoscopy and requiring blood transfusion, b) history of at least moderate ascites (on physical exam or imaging) currently treated with diuretics.
4. MELD score ≥12 and ≤20 during screening
5. Albumin ≥2.5 g/dL during screening
6. Serum creatinine ≤1.5 mg/dL during screening

Key Exclusion Criteria:

1. Evidence of severe decompensation
2. Non-cirrhotic portal hypertension
3. Child-Pugh score ≥10
4. Current use of anticoagulants that affect prothrombin time or international normalized ratio
5. ALT >3 times upper limit of normal (ULN) or AST >5 times ULN during screening
6. Initiation or discontinuation of non-selective beta blockers within 1 month of screening
7. Transjugular intrahepatic portosystemic shunt or other porto-systemic bypass procedure within 1 year of screening or previously requiring revision
8. Alpha-fetoprotein >50 ng/mL in the last year
9. History of hepatocellular carcinoma (HCC) or evidence of HCC
10. History of malignancies other than HCC, unless successfully treated with curative intent and believed to be cured
11. Prior liver transplant
12. Uncontrolled diabetes mellitus (HbA1c >9%)
13. Change in diabetes medications or vitamin E within 3 months of screening
14. Restrictive bariatric surgery or bariatric device within 1 year of screening or prior malabsorptive bariatric surgery
15. Symptoms of biliary colic unless resolved following cholecystectomy
16. History of significant alcohol consumption within the past 5 years
17. Current use of medications that are considered inhibitors of organic anion transporting polypeptide OATP1B1 and OATP1B3 transporters
18. Prolongation of screening (pre-treatment) QTcF interval of >500 msecs, or history or presence of clinically concerning cardiac arrhythmias
19. Significant systemic or major illness other than liver disease
20. Human immunodeficiency virus infection
21. Use of alcohol, controlled substances (including inhaled or injected drugs), or non-prescribed use of prescription drugs within 1 year of screening to the point of interfering with the subject's ability to comply with study procedures and study drug administration in the investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of the effect of emricasan on improving event-free survival relative to placebo, based on a composite clinical endpoint | Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks)

SECONDARY OUTCOMES:
Improvement in MELD score | Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks)
  The effect of emricasan on improving MELD score relative to placebo
Improvement in Child-Pugh scores | Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks)
  The effect of emricasan on improving the Child-Pugh score relative to placebo
Reduction of the proportion of subjects with MELD score progression | Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks)
  The effect of emricasan on reducing the proportion of patients with MELD score progression (≥4 point increase at any study visit) relative to placebo
Decrease in new decompensation events | Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks)
  The effect of emricasan on decreasing new decompensation events relative to placebo
Decrease in liver transplantation rates | Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks)
  The effect of emricasan on decreasing liver transplantation rates (in association with MELD score ≥25) relative to placebo
Decrease in all-cause and liver specific mortality | Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks)
  The effect of emricasan on decreasing all-cause and liver specific mortality relative to placebo
Improvement in health-related quality of life (QOL) as measured by Short Form-36 | Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks)
Improvement in liver metabolic function as measured by Methacetin Breath Test (MBT) | Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Chan, MD, Study Director — Conatus Pharmaceuticals Inc.
Locations (76):
- United States (76):
  - The Institute for Liver Health, Chandler, Arizona
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Arizona Liver Research Institute, Tucson, Arizona
  - University of California, San Francisco-Fresno, Fresno, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA Pfleger Liver Institute, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Stanford University, Redwood City, California
  - Inland Empire Liver Foundation, Rialto, California
  - UC Davis GI/Hepatology Clinical Trials Unit, Sacramento, California
  - Scripps Clinic - Torrey Pines, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Peak Enterology Associates, Colorado Springs, Colorado
  - West Haven VA Medical Center, West Haven, Connecticut
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Schiff Center for Liver Disease/University of Miami, Miami, Florida
  - Florida Hospital Transplant Institute, Orlando, Florida
  - IMIC Inc., Palmetto Bay, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Transplant Institute, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Aquiant Research, Albany, Indiana
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics/ Internal Medicine, Iowa City, Iowa
  - Delta Research Partners, Bastrop, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center (WRNMMC), Bethesda, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Division of Digestive Diseases, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Northwell Health Inc., Sandra Atlas Bass Center for Liver Diseases., Manhasset, New York
  - NYU Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center - Center for Liver Disease and Transplantation, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Carolinas Healthcare System, Center for Liver Disease, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - UC Health/ UCPC LLC, Cincinnati, Ohio
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - GHS Gastroenterology and Liver Center, Greenville, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Methodist Health System Clinical Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor Scott & White Research Institute, Fort Worth, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - American Research Corporation at the Texas Liver Institue, San Antonio, Texas
  - Methodist Specialty & Transplant Hospital, San Antonio, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Emeritas Research Group LLC, Leesburg, Virginia
  - Banner University Medical Center - Phoenix Transplant Institute, Newport News, Virginia
  - Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
  - University of Washington Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frenette C, Kayali Z, Mena E, Mantry PS, Lucas KJ, Neff G, Rodriguez M, Thuluvath PJ, Weinberg E, Bhandari BR, Robinson J, Wedick N, Chan JL, Hagerty DT, Kowdley KV; IDN-6556-17 Study Investigators. Emricasan to prevent new decompensation in patients with NASH-related decompensated cirrhosis. J Hepatol. 2021 Feb;74(2):274-282. doi: 10.1016/j.jhep.2020.09.029. Epub 2020 Oct 8. PMID 33038432